CLINICAL TRIAL: NCT03838120
Title: Determination of Minimum Effective Volume of Local Anesthetic in Patients Undergoing Ultrasound-Guided Infraclavicular Approach for Brachial Plexus Blockade
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: AnkaranTRH1
Record Dates: First submitted 2019-02-10; First posted 2019-02-12 (Actual); Last update posted 2021-10-27 (Actual); Status verified 2019-02

CONDITIONS: Underdosing of Local Anesthetics; Anesthetics, Local; Peripheral Nervous System Agents; Physiological Effects of Drugs
Keywords: Ultrasound; Minimum; Infraclavicular block

STUDY DESIGN:
Intervention Model Description: A total of 48 ASA I-II patients underwent upper limb surgery operation by administering USG guided-infraclavicular blockage were included in the study. brachial plexus were seen and the minimum effective LA volume was investigated starting with total 30 ml of %0.5 bupivacain. After accomplishing the blockage, volume was decreased 2ml. Block administration time, block onset times, anesthesia times and time to first analgesic requirement were recorded.
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bupivacaine 0,5% Single arm study (Other): Bupivacaine 0,5% Single arm study
  Interventions: Other: Procedure/Surgery: bupivakain % 0,5

INTERVENTIONS:
Other: Procedure/Surgery: bupivakain % 0,5 — In this study, 5 patients were included in each volume group and at least 3 applications out of 5 had to be successful to consider the volume to be sufficient. After a successful group, the volume was reduced by 2 ml's and the same procedure was followed until a final group with unsuccessful anesthesia was found (≤2 successful blockades). The study was ended at this point and MEV was determined as the volume used in the last successful group. The researcher which determined the success of blockade was blinded to the study protocol. BMI, ASA Score, Successful blockade onset time Regression time of sensorial blockade Regression time of motor blockade Time of first additional analgesic requirement

SUMMARY:
Peripheral nerve blocks with use of USG allowed visualisation of the structures and nerves and made the block administrations safe, quick and comfortable. However there are few publications concerning the minimum local anesthetic volume capable of providing blocks. In this study the investigastors aimed to find Minimum Effective Volume Of Local Anesthetic For Ultrasound-Guided İnfraclavicular Approach for Brachial Plexus Blockade in upper limb operations.

DETAILED DESCRIPTION:
This study was planned as a controlled, double-blind, single center study. Patients between 18-70 years of age who were determined as ASA I-III and underwent upper limb surgery from November 2015 to November 2016 and provided informed consent, were included in the study. Patients who had any of the following conditions were excluded: ASA risk score of IV or V, serious cardiac, respiratory, hepatic or renal comorbidities, mental disorder, coagulopathy, pregnancy, local anesthetic allergy, neuromuscular and/or neurological disease, and infection at the site of injection field of application. Patients who were unwilling to participate were also excluded. Randomization was done according to the time of patient referral with the sealed envelope system. Ethical approval was obtained from Ankara University Clinical Research Ethic Committee. All patients providedgave informed consent.

All procedures were performed by the same physician (S.B). In each patient, routine anesthesia monitoring was established and patients were administeredgiven 0.03 mg/kg midazolam and 1µg/kg of fentanyl for sedation. Field of applicationThe site of injection was properly prepared according to asepsis and antisepsis guidelines.

The infraclavicular blockade was performed according to the lateral sagittal infraclavicular block (LSIB) technique reported by Klaastad et al. [8]. The technique was modified to include ultrasound guidance, which was performed with a 6-12 mHz lineer ultrasound probe. The infraclavicular blockade was performed according to the lateral sagittal infraclavicular block (LSIB) technique reported by Klaastad et al. [8]. The technique was modified to include ultrasound guidance, which was performed with a 6-12 mHz lineer ultrasound probe. During the procedure, the patient was in the supine position with the head turned away from the application sidewith the head turned away from the application side and the shoulder was relaxed. The arm on the operative side undergoing surgery was slightly abducted, the elbow was flexed 90° and placed on the body of the patient. The anesthesiologist performing the procedure was positioned beside the head of the patient. The US probe was placed 1 cm inferior to the point of intersection between the clavicula and coracoid process on the sagittal axis. The in-plane technique was used during the procedure and the needle was visualized at all times. In order to obtain appropriate spread, the local anesthetic (0.5% [5 mg/ml] bupivacaine) was applied in a U shape from 3 to 11 o'clock around the axillary artery. U-shape distribution was achieved with (iğne pozisyonu yazılmalı); however, if distribution could not be achieved, the needle was repositioned when necessary.

The order of surgery was decided in a first come-first serve manner and Tthe volume of local anesthetic was reduced from a starting dose of 30 ml's in the first group. Five patients were included in each volume group and at least 3 applications out of 5 had to be successful to consider the volume to be sufficient. If the previous group's anesthesia was deemed as successful, the anesthesiologist reduced the dose by 2 ml's every 5 patients. When the anesthesia of a group of patients was determined to be unsuccessful (≤2 successful blockageblockades) the study was ended (Figure 1).

The researcher which determined whetherif the blockade was successful (N.A.E) was blinded to the study protocol. Sensorial and motor block measurements were used to determine blockade success. In the evaluation of sensorial blockade, touch and cold sensation tests were used to evaluate each region innervated by axillary, musculocutaneous, median, radial, and ulnar nerves. Touch sensation was evaluated with the cotton wool test and cold sensation was evaluated with ice packs. Evaluation was performed by comparing each region with the corresponding contralateral region. A score of 0 meant no blockade, 1 meant analgesia (touch sensation present, heat sensation absent), and 2 meant complete blockade of that specific region.

Motor blockade was graded on a 3-point scale; 0= no blockade, 1= partial motor blockade, 2= complete motor blockade. In this evaluation, muscles innervated by the axillary, musculocutaneous, median, radial, and ulnar nerves were each tested for motor response. The lack of movement was accepted to show complete blockade, slight movements were accepted to show partial motor blockade (initiation of motor blockade), and normal movements were considered as absence of motor blockade.

Evaluation was performed every 5 minutes during the first 60 minutes. The maximum total score for sensorial and motor blockade was 2016. During evaluation, the anesthesia and blockageblockade was accepted to be unsuccessful if this score dropped below 12. Furthermore, a sensorial blockade score of at least 97 from the possible 108 was accepted to be a requirement for successful blockade.

If unsuccessful blockade was determined during the first 60 minutes of the procedure, LMA anesthesia was applied to the patient (all applications were routine procedures and were performed with the only long-acting local anesthetic available in our hospital, 0.5% bupivacaine).

The initiation of motor and sensorial blockade was accepted as the time at which Bromage scale score changed from 0 to 1 and. tThe time of regression was accepted as the time at which score dropped below 1 for each region. The post-operative pain of patients was evaluated via the visual analogue scale (VAS) aton post-op 2, 4, 8, 12, 16, and 24 hours. Assessment of VAS was made with a 10 cm ruler with numbers from 0 to 10. The requirement for additional analgesic was accepted as the time at which VAS score increased above 4. Surgery duration, patient satisfaction and surgeon satisfaction were evaluated and measured as very good, good, moderate, and poor.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 18-70 years of age who were determined as ASA I-III and underwent upper limb surgery from November 2015 to November 2016 and provided informed consent, were included in the study.

Exclusion Criteria:

* Patients who had any of the following conditions were excluded: ASA risk score of IV or V, serious cardiac, respiratory, hepatic or renal comorbidities, mental disorder, coagulopathy, pregnancy, local anesthetic allergy, neuromuscular and/or neurological disease, and infection at the site of injection. Patients who were unwilling to participate were also excluded

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2015-11-01 (Actual); Primary Completion 2016-04-01 (Actual); Study Completion 2016-11-01 (Actual)

PRIMARY OUTCOMES:
minimum effective volume | A blinded Assistant assess sensory and motor blockade in a 5-min intervals up to 60 minutes.
  Determining the minimum effective volume of bupivacaine 0,5% for successful ultrasound guided infraclavicular brachial plexus block for upper limb surgery

SECONDARY OUTCOMES:
Successful blockade onset time | A blinded Assistant assess sensory and motor blockade in a 5-min intervals up to 60 minutes.
  Sensorial and motor block measurements were used to determine blockade success.
Regression time of sensorial blockade | post-op 2, 4, 8, 12, 16, and 24 hours.
  The initiation of motor and sensorial blockade was accepted as the time at which Bromage scale score changed from 0 to 1 and the time of regression was accepted as the time at which score dropped below 1 for each region
Regression time of motor blockade | post-op 2, 4, 8, 12, 16, and 24 hours.
  The initiation of motor and sensorial blockade was accepted as the time at which Bromage scale score changed from 0 to 1 and the time of regression was accepted as the time at which score dropped below 1 for each region
Time of first additional analgesic requirement | The post-operative pain of patients was evaluated via the visual analogue scale (VAS) at post-op 2, 4, 8, 12, 16, and 24 hours
  The requirement for additional analgesic was accepted as the time at which VAS score increased above 4hours

IPD SHARING:
Plan to Share IPD: Undecided